CLINICAL TRIAL: NCT01501071
Title: Esophageal Calibration With Soft Orogastric Tube During Laparoscopic Fundoplication Reduces Postoperative Transient Dysphagia
Brief Title: Esophageal Calibration During Laparoscopic Fundoplication Reduces Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nurullah Bulbuller, Clinical director, Antalya Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2011-12-27; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Dysphagia
Keywords: Laparoscopic Nissen fundoplication; Esophageal calibration; Postoperative dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- esophageal calibration (Experimental): Esophageal calibration tube was applied to this group of patients during laparoscopic Nissen fundoplication operation
  Interventions: Device: Esophageal calibration tube
- Control (No Intervention): Standard Laparoscopic Nissen fundoplication without esophageal calibration

INTERVENTIONS:
Device: Esophageal calibration tube — An orogastric calibration tube is inserted during laparoscopic Nissen fundoplication in order to secure a certain esophageal lumen for reducing postoperative dysphagia
  Other Names: A.M.I.Gastric tube code: AGB 355
  Arms: esophageal calibration

SUMMARY:
Gastro esophageal reflux is the most common benign disease of the esophagus and Laparoscopic Nissen fundoplication became the standard surgical treatment of this disease. Although being almost transient postoperative dysphagia is still a common complaint following this procedure. The aim of this study is to investigate the effect of inserting a soft structured and blunt mounted 39 F orogastric tube to postoperative dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* Grade 3 or more esophagitis
* Hiatal hernia larger than 3 centimeters
* Acide suppression therapy history longer than 2 years

Exclusion Criteria:

* Story of endoscopic mucosal resection for Barret's mucosa

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
dysphagia severity score | one year
  This score system is used to assess the severity of dysphagia

CONTACTS AND LOCATIONS:
Overall Officials: Nurullah Bulbuller, MD, Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Department of 2nd General Surgery, Antalya, Turkey (Türkiye)

REFERENCES:
- [Background] Nebel OT, Fornes MF, Castell DO. Symptomatic gastroesophageal reflux: incidence and precipitating factors. Am J Dig Dis. 1976 Nov;21(11):953-6. doi: 10.1007/BF01071906. PMID 984016
- [Background] Ronkainen J, Aro P, Storskrubb T, Lind T, Bolling-Sternevald E, Junghard O, Talley NJ, Agreus L. Gastro-oesophageal reflux symptoms and health-related quality of life in the adult general population--the Kalixanda study. Aliment Pharmacol Ther. 2006 Jun 15;23(12):1725-33. doi: 10.1111/j.1365-2036.2006.02952.x. PMID 16817916
- [Background] Rattner DW. Measuring improved quality of life after laparoscopic Nissen fundoplication. Surgery. 2000 Mar;127(3):258-63. doi: 10.1067/msy.2000.103881. PMID 10715979
- [Background] Terry M, Smith CD, Branum GD, Galloway K, Waring JP, Hunter JG. Outcomes of laparoscopic fundoplication for gastroesophageal reflux disease and paraesophageal hernia. Surg Endosc. 2001 Jul;15(7):691-9. doi: 10.1007/s004640080144. Epub 2001 May 7. PMID 11591970
- [Background] Pessaux P, Arnaud JP, Delattre JF, Meyer C, Baulieux J, Mosnier H. Laparoscopic antireflux surgery: five-year results and beyond in 1340 patients. Arch Surg. 2005 Oct;140(10):946-51. doi: 10.1001/archsurg.140.10.946. PMID 16230543
- [Background] Lafullarde T, Watson DI, Jamieson GG, Myers JC, Game PA, Devitt PG. Laparoscopic Nissen fundoplication: five-year results and beyond. Arch Surg. 2001 Feb;136(2):180-4. doi: 10.1001/archsurg.136.2.180. PMID 11177138
- [Background] Gotley DC, Smithers BM, Rhodes M, Menzies B, Branicki FJ, Nathanson L. Laparoscopic Nissen fundoplication--200 consecutive cases. Gut. 1996 Apr;38(4):487-91. doi: 10.1136/gut.38.4.487. PMID 8707074
- [Background] Watson DI, Pike GK, Baigrie RJ, Mathew G, Devitt PG, Britten-Jones R, Jamieson GG. Prospective double-blind randomized trial of laparoscopic Nissen fundoplication with division and without division of short gastric vessels. Ann Surg. 1997 Nov;226(5):642-52. doi: 10.1097/00000658-199711000-00009. PMID 9389398
- [Background] Hunter JG, Swanstrom L, Waring JP. Dysphagia after laparoscopic antireflux surgery. The impact of operative technique. Ann Surg. 1996 Jul;224(1):51-7. doi: 10.1097/00000658-199607000-00008. PMID 8678618
- [Background] Patterson EJ, Herron DM, Hansen PD, Ramzi N, Standage BA, Swanstrom LL. Effect of an esophageal bougie on the incidence of dysphagia following nissen fundoplication: a prospective, blinded, randomized clinical trial. Arch Surg. 2000 Sep;135(9):1055-61; discussion 1061-2. doi: 10.1001/archsurg.135.9.1055. PMID 10982510
- [Background] Richardson WS, Hunter JG. Laparoscopic floppy Nissen fundoplication. Am J Surg. 1999 Feb;177(2):155-7. doi: 10.1016/s0002-9610(98)00324-9. PMID 10204561
- [Background] Schauer PR, Meyers WC, Eubanks S, Norem RF, Franklin M, Pappas TN. Mechanisms of gastric and esophageal perforations during laparoscopic Nissen fundoplication. Ann Surg. 1996 Jan;223(1):43-52. doi: 10.1097/00000658-199601000-00007. PMID 8554418
- [Background] Lowham AS, Filipi CJ, Hinder RA, Swanstrom LL, Stalter K, dePaula A, Hunter JG, Buglewicz TG, Haake K. Mechanisms and avoidance of esophageal perforation by anesthesia personnel during laparoscopic foregut surgery. Surg Endosc. 1996 Oct;10(10):979-82. doi: 10.1007/s004649900218. PMID 8864089
- [Background] Rantanen TK, Salo JA, Salminen JT, Kellokumpu IH. Functional outcome after laparoscopic or open Nissen fundoplication: a follow-up study. Arch Surg. 1999 Mar;134(3):240-4. doi: 10.1001/archsurg.134.3.240. PMID 10088561
- [Background] Somasekar K, Morris-Stiff G, Al-Madfai H, Barton K, Hassn A. Is a bougie required for the performance of the fundal wrap during laparoscopic Nissen fundoplication? Surg Endosc. 2010 Feb;24(2):390-4. doi: 10.1007/s00464-009-0592-2. Epub 2009 Jun 24. PMID 19551431
- [Background] DeMeester TR, Bonavina L, Albertucci M. Nissen fundoplication for gastroesophageal reflux disease. Evaluation of primary repair in 100 consecutive patients. Ann Surg. 1986 Jul;204(1):9-20. doi: 10.1097/00000658-198607000-00002. PMID 3729589
- [Background] Mathavan VK, Yuh JN, Marks JM. Long-term evaluation of patients undergoing laparoscopic antireflux surgery without bougie placement. J Laparoendosc Adv Surg Tech A. 2009 Feb;19(1):7-12. doi: 10.1089/lap.2007.0135. PMID 18973468